CLINICAL TRIAL: NCT03911076
Title: A Randomized Double-Blind, Placebo-controlled Phase II Trial With Safety Run-In of Intramuscular pNGVL4a-Sig/E7(Detox)/HSP70 and TA-CIN for the Treatment of Patients With HPV16+ Atypical Squamous Cells of Undetermined Significance (ASC-US) or Cannot Exclude High Grade SIL (ASC-H) Cytology or Low-grade Squamous Intraepithelial Lesion (LSIL)
Brief Title: Phase II Study of Treatment for HPV16+ ASC-US, ASC-H and LSIL
Acronym: PVX2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment/funding
Sponsor: PapiVax Biotech, Inc. (Other)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVX2TACIN17368
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: ASC-US; ASC-H; LSIL
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix

STUDY DESIGN:
Intervention Model Description: Safety run-in followed by randomized double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Safety run-in is open label (no control), followed by randomized double-blind, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PVX-2 (Experimental): Prime: 3 mg pNGVL4a-Sig/E7(detox)/HSP70 DNA Boost: 0.1 mg TA-CIN protein
  Interventions: Biological: PVX-2
- Placebo (Placebo Comparator): Prime: PBS (Phosphate Buffered Saline) Boost: PGC (Phosphate Glycine Cysteine Buffer)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PVX-2 — pNGVL4a-Sig/E7(detox)/HSP70 (pBI-1, naked DNA plasmid priming vaccine) TA-CIN (HPV16 L2E7E6 fusion protein booster vaccine)
  Arms: PVX-2
Other: Placebo — PBS and PGC
  Arms: Placebo

SUMMARY:
* To evaluate the safety and tolerability of the dual IM pNGVL4a Sig/E7(detox)/HSP70 DNA and single IM TA-CIN immunization regimen
* To evaluate the efficacy of dual IM pNGVL4a-Sig/E7(detox)/HSP70 DNA and single IM TA-CIN immunization regimen on Human Papillomavirus (HPV) 16 clearance by Month 6

DETAILED DESCRIPTION:
Patients with human papillomavirus type 16 (HPV16) infection and low-grade cervical dysplasia [low-grade squamous intraepithelial lesion (LSIL)/CIN1] or atypical squamous cells [atypical squamous cells of undetermined significance (ASC-US)/atypical squamous cells- cannot exclude high-grade squamous intraepithelial lesion (ASC-H)] require active surveillance for disease progression. A safe and effective immunotherapy to clear HPV16 is an unmet medical need. This study (NCT03911076) is a randomized double-blind, placebo-controlled phase II trial of PVX2 [vaccination twice with HPV16-targeting pNGVL4a-Sig/E7(detox)/HSP70 plasmid and once with the HPV16 L2E7E6 fusion protein "TA-CIN"] as immunotherapy for patients with HPV16+ ASC-US, ASC-H, or LSIL/CIN1. The primary objective of this cohort is to determine the safety and tolerability of PVX2 in three monthly immunizations. Subjects are confirmed to have HPV16 infection and LSIL/CIN1, ASC-US, or ASC-H. Adverse events are evaluated using Common Terminology Criteria for Adverse Events v5.0. HPV typing by HPV16 18/45 Aptima Assay is performed at baseline, month 6, and month 12, with simultaneous cytology analysis. Cervical biopsies and endocervical curettage are performed at baseline and month 6. In a safety run-in cohort 12 eligible patients are enrolled prior to the randomized phase.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects age 25-70 years with confirmation of ASC-US, ASC-H, or LSIL by liquid-based cytology
2. HIV uninfected
3. Patients whose cytologic specimen is HPV16+ by Aptima HPV 16 18/45 Genotype Assay
4. Body Mass Index ≤ 32 kg/m2
5. Hepatitis B surface antigen negative
6. Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV positive
7. Patients who are able and willing to comply with all study procedures and voluntarily sign an informed consent form, and with anticipated availability for the planned follow-up period of one year
8. Patients who are of childbearing potential agree to remain sexually abstinent, use methods of contraception (e.g. oral contraception, barrier methods, spermicide, intrauterine device (IUD)), or have a partner who is sterile (i.e., vasectomy) through 6 months.
9. Patients must have adequate organ function at the time of enrollment as defined by the following parameters: white blood cell count >3,000/mcL; lymphocyte number >500/mcL; absolute neutrophil count >1,000/mcL; platelets >90,000/mcL; hemoglobin >9 g/dL; total bilirubin <3 X the institutional limit of normal; aspartate aminotransferase (AST [SGOT]) / alanine aminotransferase (ALT [SGPT]) <3 X the institutional limit of normal; creatinine <2.5X the institutional limit of normal.
10. Histologic diagnosis of <CIN2 upon screening colposcopic examination with mandatory ECC, and cervical biopsy(ies) as clinically indicated.

Exclusion Criteria:

1. Patients who are attempting pregnancy within 6 months, pregnant, or breastfeeding.
2. Patients with immunodeficiency, or treatment with immunosuppressive medications
3. Administration of any blood product within 3 months of enrollment.
4. Administration of any licensed vaccine within 2 weeks of enrollment (4weeks for measles vaccine)
5. Participation in a study with an investigational compound or device within 30 days of signing informed consent.
6. History of seizures (unless seizure free for 5 years)
7. Patients with positive serological test for human immunodeficiency virus (HIV).
8. Previous cancer history within the past 5 years.
9. Patients who have had chemotherapy, radiation, biological cancer therapy, or other investigational agents within 28 days prior to the first dose of study drug.
10. Patients who have had surgery within 28 days, excluding minor procedures (dental work, skin biopsy, etc).
11. Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing, or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Patients who have an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis).
13. Patients with a recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia, or dysgammaglobulinemia; patients who have acquired, hereditary, or congenital immunodeficiencies; patients being chronically treated with immunosuppressive drugs such as cyclosporin, adrenocorticotropic hormone (ACTH), or systemic corticosteroids
14. Previous cervical conization or LEEP procedure or previous total hysterectomy due to cervical lesions at enrollment.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with cervical cytologic diagnosis of ASC-US, ASC-H, or LSIL
Enrollment: 16 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | 12 months
  To evaluate the safety and tolerability of the dual IM pNGVL4a Sig/E7(detox)/HSP70 DNA and single IM TA-CIN immunization regimen
Percent of patients that have cleared HPV16 at Month 6 | 6 months
  To evaluate the efficacy of dual IM pNGVL4a-Sig/E7(detox)/HSP70 DNA and single IM TA-CIN immunization regimen on Human Papillomavirus (HPV) 16 clearance by Month 6

SECONDARY OUTCOMES:
Percent of patients that have cleared HPV16 at Month 12 | 12 months
  To evaluate the efficacy of dual IM pNGVL4a-Sig/E7(detox)/HSP70 DNA and single IM TA-CIN immunization regimen on maintenance of Human Papillomavirus (HPV) 16 clearance by Month 12
Percent of patients that have normal cytology at Month 6 | 6 months
  To evaluate the efficacy of dual IM pNGVL4a-Sig/E7(detox)/HSP70 DNA and single IM TA-CIN immunization regimen on regression to cytology with no evidence of intraepithelial lesion or malignancy (NILM) at Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Mark Einstein, MD, MS, Principal Investigator — Professor and Chairman, Dept. of OBS&GYN, Rutgers New Jersey Medical School, Newark, NJ 07101
Locations (6):
- United States (6):
  - Health Awareness, Inc., Port Saint Lucie, Florida
  - University Hospital, Rutgers New Jersey Medical School, Newark, New Jersey
  - Obstetrics & Gynecology Associates, Inc., Fairfield, Ohio
  - Austin Area Obstetrics, Gynecology, and Fertility, Austin, Texas
  - Corpus Christi Women's Clinic (Elligo Health Research, Inc.), Corpus Christi, Texas
  - MacArthur Medical Center, Irving, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Einstein MH, Roden RBS, Ferrall L, Akin M, Blomer A, Wu TC, Chang YN. Safety Run-in of Intramuscular pNGVL4a-Sig/E7(detox)/HSP70 DNA and TA-CIN Protein Vaccination as Treatment for HPV16+ ASC-US, ASC-H, or LSIL/CIN1. Cancer Prev Res (Phila). 2023 Apr 3;16(4):219-227. doi: 10.1158/1940-6207.CAPR-22-0413. PMID 36607735
- See also: Study report — https://pubmed.ncbi.nlm.nih.gov/36607735/